CLINICAL TRIAL: NCT00417079
Title: A Randomized, Open Label Multi-Center Study of XRP6258 at 25 mg/m^2 in Combination With Prednisone Every 3 Weeks Compared to Mitoxantrone in Combination With Prednisone For The Treatment of Hormone Refractory Metastatic Prostate Cancer Previously Treated With A Taxotere®-Containing Regimen
Brief Title: XRP6258 Plus Prednisone Compared to Mitoxantrone Plus Prednisone in Hormone Refractory Metastatic Prostate Cancer
Acronym: TROPIC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: International Clinical Development Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EFC6193
Record Dates: First submitted 2006-12-28; First posted 2006-12-29 (Estimated); Results first posted 2010-12-23 (Estimated); Last update posted 2011-03-10 (Estimated); Status verified 2011-03

CONDITIONS: Neoplasms; Prostatic Neoplasms
Keywords: Cancer; Prostate
MeSH Terms: conditions — Neoplasms; Prostatic Neoplasms | interventions — cabazitaxel; XRP6258; Mitoxantrone; Prednisone

ARMS (2):
- Mitoxantrone + Prednisone (Active Comparator): Mitoxantrone + Prednisone
  Interventions: Drug: mitoxantrone; Drug: prednisone
- Cabazitaxel + Prednisone (Experimental): Cabazitaxel + Prednisone
  Interventions: Drug: cabazitaxel (XRP6258) (RPR116258); Drug: prednisone

INTERVENTIONS:
Drug: cabazitaxel (XRP6258) (RPR116258) — 25 mg/m^2 administered by intravenous (IV) route over 1 hour on day 1 of each 21-day cycle
  Other Names: Jevtana
  Arms: Cabazitaxel + Prednisone
Drug: mitoxantrone — 12 mg/m^2 administered by intravenous (IV) route over 15-30 minutes on day 1 of each 21-day cycle
  Arms: Mitoxantrone + Prednisone
Drug: prednisone — 10 mg daily administered by oral route

SUMMARY:
This is a randomized, open-label, multi-center study comparing the safety and efficacy of XRP6258 plus prednisone to mitoxantrone plus prednisone in the treatment of hormone refractory metastatic prostate cancer previously treated with a Taxotere®-containing regimen. The primary objective is overall survival. Secondary objectives include progression free survival, overall response rate, prostate-specific antigen (PSA) response/progression, pain response/progression, overall safety, and pharmacokinetics. Patients will be treated until disease progression, death, unacceptable toxicity, or for a maximum of 10 cycles. Patients will have long-term follow-up for a maximum of up to 2 years.

ELIGIBILITY:
Inclusion Criteria

1. Histologically or cytologically confirmed adenocarcinoma of the prostate that is refractory to hormone therapy and previously treated with a Taxotere®-containing regimen.
2. Documented progression of disease (demonstrating at least one visceral or soft tissue metastatic lesion, including a new lesion). Patients with non-measurable disease must have documented rising prostate-specific antigen (PSA) levels or appearance of new lesion.
3. Surgical or hormone-induced castration
4. Life expectancy > 2 months
5. Eastern Cooperative Oncology Group (ECOG) performance status 0 - 2

Exclusion criteria

1. Previous treatment with mitoxantrone
2. Previous treatment with <225 mg/m^2 cumulative dose of Taxotere (or docetaxel)
3. Prior radiotherapy to ≥ 40% of bone marrow
4. Surgery, radiation, chemotherapy, or other anti-cancer therapy within 4 weeks prior to enrollment in the study
5. Other prior malignancy, except for adequately treated superficial basal cell skin cancer, or any other cancer from which the patient has been disease-free for less than 5 years
6. Known brain or leptomeningeal involvement
7. Other concurrent serious illness or medical conditions
8. Inadequate organ function evidenced by unacceptable laboratory results

The investigator will evaluate whether there are other reasons why a patient may not participate.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 755 (Actual)
Dates: Start 2007-01; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ICD, Study Director — Sanofi
Locations (26):
- sanofi-aventis US, Bridgewater, New Jersey, United States
- sanofi-aventis Argentina, Buenos Aires, Argentina
- sanofi-aventis Belgium, Diegem, Belgium
- sanofi-aventis Brazil, São Paulo, Brazil
- sanofi-aventis Canada, Laval, Quebec, Canada
- sanofi-aventis Chile, Santiago, Chile
- sanofi-aventis Czech Republic, Prague, Czechia
- sanofi-aventis Denmark, Hørsholm, Denmark
- sanofi-aventis Finland, Helsinki, Finland
- sanofi-aventis France, Paris, France
- sanofi-aventis Germany, Berlin, Germany
- Sanofi-Aventis Hungaria, Budapest, Hungary
- sanofi-aventis India, Mumbai, India
- sanofi-aventis Italy, Milan, Italy
- sanofi-aventis Mexico, México, Mexico
- sanofi-aventis Netherlands, Gouda, Netherlands
- sanofi-aventis Russia, Moscow, Russia
- sanofi-aventis Singapore, Singapore, Singapore
- sanofi-aventis Slovakia, Bratislava, Slovakia
- sanofi-aventis South Africa, Midrand, South Africa
- sanofi-aventis South Korea, Seoul, South Korea
- sanofi-aventis Spain, Barcelona, Spain
- sanofi-aventis Sweden, Bromma, Sweden
- sanofi-aventis Taiwan, Taipei, Taiwan
- sanofi-aventis Turkey, Istanbul, Turkey (Türkiye)
- sanofi-aventis UK, Guildford, Surrey, United Kingdom

REFERENCES:
- [Derived] Lorente D, Mateo J, Templeton AJ, Zafeiriou Z, Bianchini D, Ferraldeschi R, Bahl A, Shen L, Su Z, Sartor O, de Bono JS. Baseline neutrophil-lymphocyte ratio (NLR) is associated with survival and response to treatment with second-line chemotherapy for advanced prostate cancer independent of baseline steroid use. Ann Oncol. 2015 Apr;26(4):750-755. doi: 10.1093/annonc/mdu587. Epub 2014 Dec 23. PMID 25538172
- [Derived] Bahl A, Oudard S, Tombal B, Ozguroglu M, Hansen S, Kocak I, Gravis G, Devin J, Shen L, de Bono JS, Sartor AO; TROPIC Investigators. Impact of cabazitaxel on 2-year survival and palliation of tumour-related pain in men with metastatic castration-resistant prostate cancer treated in the TROPIC trial. Ann Oncol. 2013 Sep;24(9):2402-8. doi: 10.1093/annonc/mdt194. Epub 2013 May 30. PMID 23723295
- [Derived] Pouessel D, Oudard S, Gravis G, Priou F, Shen L, Culine S. [Cabazitaxel for metastatic castration-resistant prostate cancer progressing after docetaxel treatment: the TROPIC study in France]. Bull Cancer. 2012 Jul-Aug;99(7-8):731-41. doi: 10.1684/bdc.2012.1608. French. PMID 22743148
- [Derived] de Bono JS, Oudard S, Ozguroglu M, Hansen S, Machiels JP, Kocak I, Gravis G, Bodrogi I, Mackenzie MJ, Shen L, Roessner M, Gupta S, Sartor AO; TROPIC Investigators. Prednisone plus cabazitaxel or mitoxantrone for metastatic castration-resistant prostate cancer progressing after docetaxel treatment: a randomised open-label trial. Lancet. 2010 Oct 2;376(9747):1147-54. doi: 10.1016/S0140-6736(10)61389-X. PMID 20888992

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Multicenter study: 146 actives sites from 26 countries in Europe, USA, South America and Asia Pacific region. Study initiation date: January 2nd, 2007; study completion date/study cut off date: September 25th, 2009.
Pre-assignment Details: 165 patients signed informed consent but were not randomized and considered as screen failure.
  Intention to Treat Population (ITT or randomized patients): 755 patients (377 mitoxantrone, 378 cabazitaxel).
  Safety population (treated patients): 742 patients (371 mitoxantrone, 371 cabazitaxel) (Patients not treated: 6 mitoxantrone, 7 cabazitaxel).
Groups:
- Mitoxantrone + Prednisone: mitoxantrone 12 mg/m^2 (Day 1) by intravenous (IV) every 3 weeks, and prednisone 10 mg orally given daily
- Cabazitaxel + Prednisone: cabazitaxel 25 mg/m^2 (Day 1) by intravenous (IV) every 3 weeks, and prednisone 10 mg orally given daily
Period: Overall Study
Arm/Group | Mitoxantrone + Prednisone | Cabazitaxel + Prednisone
Started | 377 (Randomized patients) | 378 (Randomized patients)
Completed | 46 (Randomized patients) | 105 (Randomized patients)
Not Completed | 331 | 273
Not completed — Disease progression | 267 | 180
Not completed — Adverse Event | 32 | 67
Not completed — Non-compliance to protocol | 0 | 1
Not completed — Lost to Follow-up | 2 | 0
Not completed — Withdrawal by Subject | 17 | 8
Not completed — Not treated | 6 | 7
Not completed — Screened failure | 2 | 1
Not completed — Investigator's decision | 1 | 4
Not completed — Non-confirmed Disease progression | 1 | 1
Not completed — Clinical deterioration | 1 | 0
Not completed — Screening error | 2 | 1
Not completed — Withdrawal by subject's family | 0 | 1
Not completed — Patient unable to come to the clinic | 0 | 1
Not completed — abnormal liver function tests | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mitoxantrone + Prednisone | Cabazitaxel + Prednisone | Total
Number analyzed (Participants) | 377 | 378 | 755
Age Continuous [Median (Full Range); unit: years] | 67.0 [47 to 89] | 68.0 [46 to 92] | 67 [46 to 92]
Sex/Gender, Customized [Number; unit: participants]
  Male | 377 | 378 | 755
Region of Enrollment [Number; unit: participants]
  United States | 106 | 97 | 203
  Taiwan | 4 | 7 | 11
  Slovakia | 1 | 1 | 2
  Spain | 10 | 9 | 19
  Chile | 9 | 12 | 21
  Russian Federation | 6 | 4 | 10
  Italy | 17 | 18 | 35
  India | 11 | 9 | 20
  France | 44 | 46 | 90
  Denmark | 19 | 26 | 45
  South Africa | 7 | 9 | 16
  Netherlands | 8 | 9 | 17
  Korea, Republic of | 8 | 7 | 15
  Finland | 4 | 1 | 5
  Turkey | 17 | 19 | 36
  United Kingdom | 17 | 20 | 37
  Hungary | 8 | 7 | 15
  Czech Republic | 10 | 12 | 22
  Mexico | 2 | 3 | 5
  Canada | 16 | 16 | 32
  Argentina | 7 | 3 | 10
  Brazil | 7 | 4 | 11
  Belgium | 16 | 15 | 31
  Singapore | 6 | 3 | 9
  Germany | 6 | 11 | 17
  Sweden | 11 | 10 | 21
Eastern Cooperative Oncology Group (ECOG) Performance Status [Number; unit: Participants]
  0 - Fully Active | 120 | 141 | 261
  1 - Ambulatory, Restricted Activity | 224 | 209 | 433
  2 - Ambulatory, No Work Activities | 33 | 28 | 61
Prostatic Specific Antigen PSA [Median (Full Range); unit: ng/mL] | 127.5 [2 to 11220] | 143.9 [2 to 7842] | 135.00 [2 to 11220]
Measurable disease [Number; unit: Participants] — Measurability of the disease per Response Evaluation Criteria in Solid Tumors (RECIST) criteria:
  Patients with measurable disease have at least one visceral or soft tissue metastatic lesion (including new lesion).
  Patient with non-measurable disease have documented rising PSA levels or appearance of new lesion.
  Participants
    Measurable disease | 204 | 201 | 405
    Not Measurable disease | 173 | 177 | 350
Extent of disease [Number; unit: Participants] — Extent of the disease at screening stage:
  * Metastatic: bone or visceral metastases.
  * Locoregional recurrence includes local recurrent tumor at the primary site, along the draining lymphatic channels, or within the draining lymphatic nodal basin.
  Participants
    Metastatic | 356 | 364 | 720
    Locoregional Recurrence | 20 | 14 | 34
    Missing | 1 | 0 | 1
Tumor Location: number of sites involved [Number; unit: Participants]
  1 | 134 | 146 | 280
  2 | 117 | 112 | 229
  3 | 78 | 73 | 151
  4 or more | 43 | 44 | 87
  Missing | 5 | 3 | 8

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Overall survival was defined as the time interval from the date of randomization to the date of death due to any cause.
  In the absence of confirmation of death, the survival time was censored at the last date patient was known to be alive or at the cut-off date, whichever had come first.
Time Frame: From the date of randomization up to 104 weeks (study cut-off)
Population: Analysis was performed on the intention To Treat (ITT) population. The ITT population is composed of all randomized patients (i.e. patients assigned to a treatment group by the randomization, regardless of whether patients received any study drug or received a different study drug from which they were randomized).
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Mitoxantrone + Prednisone | Cabazitaxel + Prednisone
Number analyzed (Participants) | 377 | 378
Months | 12.7 [11.6 to 13.7] | 15.1 [14.1 to 16.3]
Statistical Analysis 1: Comparison: Mitoxantrone + Prednisone vs Cabazitaxel + Prednisone; The study required an estimated sample size of 720 patients (360 per arm) in order to detect a 25% reduction in the hazard ratio for death in the cabazitaxel group relative to the mitoxantrone group with 90% power. The final analysis was planned for when 511 deaths had occurred; Test type: Superiority or Other; p < 0.0001, Log Rank — A 2-sided significance level of 0.0452 was used for the final analysis based on an interim analysis performed after 307 events with an adjusted significance level of 0.016 based on the O'Brien-Fleming type 1 error spending function; Analysis was performed by using a log-rank comparisons stratified according to disease measurability and ECOG performance status (0-1 versus 2)

2. Secondary Outcome: Time to Progression Free Survival (PFS)
Description: Progression free survival was defined as a composite endpoint evaluated from the date of randomization to the date of tumor progression, PSA progression, pain progression, or death due to any cause, whichever occurred first
Time Frame: From the date of randomization up to 104 weeks (study cut-off)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Mitoxantrone + Prednisone | Cabazitaxel + Prednisone
Number analyzed (Participants) | 377 | 378
Months | 1.4 [1.4 to 1.7] | 2.8 [2.4 to 3.0]
Statistical Analysis 1: Comparison: Mitoxantrone + Prednisone vs Cabazitaxel + Prednisone; Test type: Superiority or Other; p < 0.0001, Log Rank

3. Secondary Outcome: Overall Tumor Response
Description: Tumor Overall Response Rate (ORR) (only in patients with measurable disease):
  Objective responses (Complete Response and Partial Response) for measurable disease as assessed by investigators according to RECIST criteria.
  Complete Response (CR) is defined as: Disappearance of all target lesions. Partial Response (PR) is defined as: At least a 30% decrease in the sum of longest diameter (LD) of target lesions taking as reference baseline sum LD.
  Confirmation of objective responses will be performed by repeat tumor imaging (CT scans, MRI, bone scans) after the first documentation of response.
Time Frame: From the date of randomization up to 104 weeks (study cut-off)
Population: Tumor response rate was evaluated only for patients, in the Intention-To-Treat (ITT) population, with measurable disease by Response Evaluation Criteria in Solid Tumor (RECIST).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Mitoxantrone + Prednisone | Cabazitaxel + Prednisone
Number analyzed (Participants) | 204 | 201
percentage of participants | 4.4 [1.6 to 7.2] | 14.4 [9.6 to 19.3]
Statistical Analysis 1: Comparison: Mitoxantrone + Prednisone vs Cabazitaxel + Prednisone; Test type: Superiority or Other; p = 0.0005, Chi-squared

4. Secondary Outcome: Time to Tumor Progression
Description: Time to tumor progression is defined as the number of months from randomization until evidence of progressive disease (RECIST)
Time Frame: From the date of randomization up to 104 weeks (study cut-off)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Mitoxantrone + Prednisone | Cabazitaxel + Prednisone
Number analyzed (Participants) | 377 | 378
Months | 5.4 [4.7 to 6.5] | 8.8 [7.4 to 9.6]
Statistical Analysis 1: Comparison: Mitoxantrone + Prednisone vs Cabazitaxel + Prednisone; Test type: Superiority or Other; p < 0.0001, Log Rank; Log-rank comparisons stratified according to disease measurability and ECOG performance status; Cox Proportional Hazard = 0.61, 95% CI 2-sided [0.49 to 0.76] — Hazard ratio (HR) < 1 favours the cabazitaxel group and > 1 favours the mitoxantrone group

5. Secondary Outcome: Time to Prostatic Specific Antigen (PSA) Progression
Description: In PSA non-responders, progression will be defined as a 25% increase over nadir and increase in the absolute value PSA level by at least 5 ng/ml and confirmed by a second value at least 4 weeks later.
  In PSA responders and in patients not evaluable for PSA response at baseline, progression will be defined as a ≥50% increase over nadir, provided that the increase is a minimum of 5 ng/ml and confirmed by a second value at least 1 week later.
Time Frame: at screening, day 1 of every treatment cycle, up to 104 weeks (study cut-off)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Mitoxantrone + Prednisone | Cabazitaxel + Prednisone
Number analyzed (Participants) | 377 | 378
Months | 3.1 [2.2 to 4.4] | 6.4 [5.1 to 7.3]
Statistical Analysis 1: Comparison: Mitoxantrone + Prednisone vs Cabazitaxel + Prednisone; Test type: Superiority or Other; p = 0.0010, Log Rank; Log-rank comparisons stratified according to disease measurability and ECOG performance status; Cox Proportional Hazard = 0.75, 95% CI 2-sided [0.63 to 0.90] — Hazard ratio (HR) < 1 favours the cabazitaxel group and > 1 favours the mitoxantrone group

6. Secondary Outcome: PSA (Prostate-Specific Antigen) Response
Description: PSA response was defined as a ≥ 50% reduction in serum PSA, determined only for patients with a serum PSA ≥ 20ng/mL at baseline, confirmed by a repeat PSA ≥ 3 weeks later.
Time Frame: from baseline up to 104 weeks (study cut-off)
Population: Prostate Specific Antigen (PSA) response was evaluated only in patients, in the Intention-To-Treat population, with a baseline PSA >20ng/mL.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Mitoxantrone + Prednisone | Cabazitaxel + Prednisone
Number analyzed (Participants) | 325 | 329
Percentage of participants | 17.8 [13.7 to 22.0] | 39.2 [33.9 to 44.5]
Statistical Analysis 1: Comparison: Mitoxantrone + Prednisone vs Cabazitaxel + Prednisone; Test type: Superiority or Other; p = 0.0002, Chi-squared

7. Secondary Outcome: Time to Pain Progression
Description: Pain Progression is defined as an increase of ≥1 point in the median Personal Pain Intensity (PPI) from its nadir noted on 2 consecutive 3-week-apart visits or ≥25 % increase in the mean analgesic score compared with the baseline score & noted on 2 consecutive 3-week-apart visits or requirement for local palliative radiotherapy.
  Evaluation of the PPI & analgesic scores are based on the short-form McGill Pain Questionnaire which consists of 15 descriptors (11 sensory; 4 affective) which are rated on an intensity scale as 0=none (best) 1=mild 2=moderate 3=severe (worst) (TOTAL: 0=best 45=worst)
Time Frame: from baseline up to 104 weeks (study cut-off)
Population: Analysis was performed on the intention To Treat (ITT) population. Data from 265 and 279 patients in the cabazitaxel and mitoxantrone groups, respectively, were censored as a results of > 2 PPI and/or AS assessments being missed during the same week (unless a complete evaluation of ≥5 values showed pain progression).
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Mitoxantrone + Prednisone | Cabazitaxel + Prednisone
Number analyzed (Participants) | 377 | 378
Months | NA [NA to NA] — Median not reached | 11.1 [8.1 to NA] — Upper confidence interval unevaluable
Statistical Analysis 1: Comparison: Mitoxantrone + Prednisone vs Cabazitaxel + Prednisone; Test type: Superiority or Other; p = 0.5192, Log Rank; Log-rank comparisons stratified according to disease measurability and ECOG performance status; Cox Proportional Hazard = 0.91, 95% CI 2-sided [0.69 to 1.19] — Hazard ratio (HR) < 1 favours the cabazitaxel group and > 1 favours the mitoxantrone group

8. Secondary Outcome: Pain Response
Description: Pain Response was defined as a two-point or greater reduction from baseline median Present Pain Intensity (PPI) score without an increased Analgesic Score (AS) or a decrease of ≥50% in the AS without an increase in the PPI score, maintained for at least 3 weeks.
Time Frame: from baseline up to 104 weeks (study cut-off)
Population: Pain Response (applies only to patients, in the Intention-To-Treat (ITT) population, with median PPI ≥2 on McGill-Melzack scale and/or mean Analgesic Score ≥10 points at baseline)
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Mitoxantrone + Prednisone | Cabazitaxel + Prednisone
Number analyzed (Participants) | 168 | 174
Percentage of participants | 7.7 [3.7 to 11.8] | 9.2 [4.9 to 13.5]
Statistical Analysis 1: Comparison: Mitoxantrone + Prednisone vs Cabazitaxel + Prednisone; Test type: Superiority or Other; p = 0.6286, Chi-squared

ADVERSE EVENTS:
Time Frame: Adverse events are collected from the time to the first patient signed an informed consent form until 30 days after the administration of the last cycle of the study treatment to the last patient (i.e. 104 weeks).
Description: The safety analyses are performed on the safety population which includes all randomized patients who received at least part of one dose of the study drug.
Arm/Group | Mitoxantrone + Prednisone | Cabazitaxel + Prednisone
Serious Adverse Events (participants affected / at risk) | 77/371 | 145/371
Other Adverse Events (participants affected / at risk) | 323/371 | 350/371
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mitoxantrone + Prednisone (N=371) | Cabazitaxel + Prednisone (N=371)
Febrile neutropenia (Blood and lymphatic system disorders) | 4 | 25
Neutropenia (Blood and lymphatic system disorders) | 3 | 18
Leukopenia (Blood and lymphatic system disorders) | 0 | 3
Anaemia (Blood and lymphatic system disorders) | 2 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 2
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 2
Cardiac arrest (Cardiac disorders) | 0 | 2
Cardiac failure (Cardiac disorders) | 0 | 2
Ventricular fibrillation (Cardiac disorders) | 0 | 1
Cardiotoxicity (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 9
Vomiting (Gastrointestinal disorders) | 2 | 6
Abdominal pain (Gastrointestinal disorders) | 0 | 6
Constipation (Gastrointestinal disorders) | 1 | 3
Nausea (Gastrointestinal disorders) | 1 | 3
Intestinal obstruction (Gastrointestinal disorders) | 0 | 3
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 2
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1
Caecitis (Gastrointestinal disorders) | 0 | 1
Duodenal ulcer perforation (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1
Enterocolitis (Gastrointestinal disorders) | 0 | 1
Enterovesical fistula (Gastrointestinal disorders) | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 1
Mesenteric vein thrombosis (Gastrointestinal disorders) | 0 | 1
Oesophageal ulcer (Gastrointestinal disorders) | 0 | 1
Haematemesis (Gastrointestinal disorders) | 2 | 0
Pancreatic mass (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Proctalgia (Gastrointestinal disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 6
Asthenia (General disorders) | 0 | 2
Chest pain (General disorders) | 0 | 2
Disease progression (General disorders) | 11 | 1
Fatigue (General disorders) | 0 | 1
Influenza like illness (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 0 | 1
Pain (General disorders) | 0 | 1
Sudden death (General disorders) | 0 | 1
Bile duct stone (Hepatobiliary disorders) | 0 | 1
Biliary colic (Hepatobiliary disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Cholangitis (Hepatobiliary disorders) | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 0
Anaphylactic shock (Immune system disorders) | 0 | 1
Pneumonia (Infections and infestations) | 2 | 6
Urinary tract infection (Infections and infestations) | 3 | 4
Sepsis (Infections and infestations) | 0 | 4
Septic shock (Infections and infestations) | 0 | 4
Neutropenic sepsis (Infections and infestations) | 1 | 3
Infection (Infections and infestations) | 2 | 2
Neutropenic infection (Infections and infestations) | 0 | 2
Salmonellosis (Infections and infestations) | 0 | 2
Cellulitis (Infections and infestations) | 2 | 1
Urosepsis (Infections and infestations) | 2 | 1
Cystitis (Infections and infestations) | 1 | 1
Lobar pneumonia (Infections and infestations) | 1 | 1
Bacteraemia (Infections and infestations) | 0 | 1
Bronchopneumonia (Infections and infestations) | 0 | 1
Campylobacter infection (Infections and infestations) | 0 | 1
Fungal sepsis (Infections and infestations) | 0 | 1
Groin abscess (Infections and infestations) | 0 | 1
Implant site cellulitis (Infections and infestations) | 0 | 1
Oesophageal candidiasis (Infections and infestations) | 0 | 1
Pneumonia klebsiella (Infections and infestations) | 0 | 1
Urinary tract infection enterococcal (Infections and infestations) | 0 | 1
Urinary tract infection fungal (Infections and infestations) | 0 | 1
Bacterial sepsis (Infections and infestations) | 1 | 0
Febrile infection (Infections and infestations) | 1 | 0
Pneumococcal sepsis (Infections and infestations) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 2
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1
Accidental overdose (Injury, poisoning and procedural complications) | 1 | 0
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 | 0
Fracture (Injury, poisoning and procedural complications) | 1 | 0
Multiple fractures (Injury, poisoning and procedural complications) | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0
Eastern cooperative oncology group performance status worsened (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 4
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 2
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 2 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Metastatic pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Spinal cord compression (Nervous system disorders) | 3 | 4
Syncope (Nervous system disorders) | 1 | 2
Cerebral haemorrhage (Nervous system disorders) | 0 | 1
Grand mal convulsion (Nervous system disorders) | 0 | 1
Metabolic encephalopathy (Nervous system disorders) | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 0 | 1
Speech disorder (Nervous system disorders) | 0 | 1
Vith nerve paralysis (Nervous system disorders) | 0 | 1
Altered state of consciousness (Nervous system disorders) | 1 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Cranial nerve paralysis (Nervous system disorders) | 1 | 0
Epiduritis (Nervous system disorders) | 1 | 0
Peripheral motor neuropathy (Nervous system disorders) | 1 | 0
Vestibular nystagmus (Nervous system disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 3 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 1
Psychotic disorder (Psychiatric disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 3 | 10
Renal failure (Renal and urinary disorders) | 0 | 6
Renal failure acute (Renal and urinary disorders) | 0 | 5
Hydronephrosis (Renal and urinary disorders) | 1 | 4
Ureteric obstruction (Renal and urinary disorders) | 0 | 4
Urinary retention (Renal and urinary disorders) | 2 | 2
Ureteric stenosis (Renal and urinary disorders) | 1 | 1
Bladder neck obstruction (Renal and urinary disorders) | 0 | 1
Renal colic (Renal and urinary disorders) | 0 | 1
Urethral pain (Renal and urinary disorders) | 0 | 1
Urethral stenosis (Renal and urinary disorders) | 0 | 1
Urinary tract obstruction (Renal and urinary disorders) | 0 | 1
Postrenal failure (Renal and urinary disorders) | 1 | 0
Penile oedema (Reproductive system and breast disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 6 | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 2 | 2
Haematoma (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 1
Extremity necrosis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Mitoxantrone + Prednisone (N=371) | Cabazitaxel + Prednisone (N=371)
Neutropenia (Blood and lymphatic system disorders) | 38 | 66
Anaemia (Blood and lymphatic system disorders) | 18 | 38
Diarrhoea (Gastrointestinal disorders) | 39 | 170
Nausea (Gastrointestinal disorders) | 84 | 127
Vomiting (Gastrointestinal disorders) | 36 | 80
Constipation (Gastrointestinal disorders) | 56 | 73
Abdominal pain (Gastrointestinal disorders) | 13 | 38
Dyspepsia (Gastrointestinal disorders) | 6 | 25
Abdominal pain upper (Gastrointestinal disorders) | 5 | 20
Fatigue (General disorders) | 102 | 136
Asthenia (General disorders) | 46 | 76
Pyrexia (General disorders) | 22 | 40
Oedema peripheral (General disorders) | 34 | 34
Mucosal inflammation (General disorders) | 10 | 22
Pain (General disorders) | 18 | 19
Urinary tract infection (Infections and infestations) | 9 | 24
Weight decreased (Investigations) | 28 | 32
Anorexia (Metabolism and nutrition disorders) | 39 | 59
Back pain (Musculoskeletal and connective tissue disorders) | 41 | 58
Arthralgia (Musculoskeletal and connective tissue disorders) | 31 | 39
Pain in extremity (Musculoskeletal and connective tissue disorders) | 27 | 29
Muscle spasms (Musculoskeletal and connective tissue disorders) | 10 | 27
Bone pain (Musculoskeletal and connective tissue disorders) | 19 | 19
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 20 | 18
Dysgeusia (Nervous system disorders) | 15 | 41
Dizziness (Nervous system disorders) | 21 | 30
Neuropathy peripheral (Nervous system disorders) | 4 | 30
Headache (Nervous system disorders) | 19 | 28
Peripheral sensory neuropathy (Nervous system disorders) | 5 | 20
Haematuria (Renal and urinary disorders) | 13 | 58
Dysuria (Renal and urinary disorders) | 5 | 25
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 16 | 43
Cough (Respiratory, thoracic and mediastinal disorders) | 22 | 40
Alopecia (Skin and subcutaneous tissue disorders) | 18 | 37
Hypotension (Vascular disorders) | 9 | 19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication of the study will be made jointly in the name of all wholehearted collaborators. Other papers will be authored based on the contributions of the individuals to the overall study. Substudies with scientific merit which have received prior approval from the Steering Committee (SC) may be published in the names of the contributing investigators. A copy of all manuscripts will be provided to the sponsors for their review. The final decision to publish articles will be made by the SC.